CLINICAL TRIAL: NCT06546865
Title: Slim Sheath 22F Holmium Laser Enucleation of the Prostate (HoLEP) Technique vs 26 F Sheath HoLEP for Treatment of Benign Prostatic Hyperplasia (BPH): A Randomized Prospective Comparative Study
Brief Title: Slim Sheath 22F Holmium Laser Enucleation of the Prostate (HoLEP) vs 26 F Sheath HoLEP for BPH: RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thunder Bay Regional Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RP-1064
Record Dates: First submitted 2024-07-30; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 22F Sheath Size (Active Comparator): Comparator arm for procedures using 22F sheath size
  Interventions: Device: 22F Sheath Size
- 26F Sheath Size (Active Comparator): Comparator arm for procedures using 26F sheath size
  Interventions: Device: 26F Sheath Size

INTERVENTIONS:
Device: 22F Sheath Size — Participants in this group will have the 22F sheath size used in their procedure.
  Arms: 22F Sheath Size
Device: 26F Sheath Size — Participants in this group will have the 26F sheath size used in their procedure.
  Arms: 26F Sheath Size

SUMMARY:
Holmium laser enucleation of the prostate (HoLEP) is routinely performed with 24F, 26F, and 28F laser scopes. Proponents of larger caliber scopes suggest that the larger scope size allows for improved visualization, hemostasis, and operative efficiencies. Proponents of a smaller scope diameter suggest that by eliminating the need for pre-HoLEP urethral dilation to accommodate a larger scope. It has also been proposed that a smaller caliber scope is less traumatic to the urethra resulting in lower rates of bladder neck contracture and urethral stricture disease. Currently, to our knowledge, there are no level one evaluation examining scope size 22F versus 26F sheath in laser enucleation outcomes. The aim of our study is to determine if a smaller diameter scope is associated with improved laser enucleation time, post-operative recovery, rates of same-day discharge, or increasing intra-operative or postoperative complication rates

ELIGIBILITY:
Inclusion Criteria:

1. Males over 50 years of age at the time of enrollment
2. Referred to urology for refractory LUTS secondary to BPH
3. Failed medical (non-surgical) treatment
4. Prostate size on preoperative TRUS of > 80 ml
5. IPSS >15, QOL score ≥3 and Qmax <15 ml/sec
6. Written informed consent to participate in the study
7. Ability to comply with the requirements of the study procedures

Exclusion Criteria:

1. Previous surgical treatment for BPH
2. History of prostate cancer
3. Prostate size < 80 mL
4. History of urethral stenosis or its management
5. Known or suspected neurogenic bladder
6. Participants with active urinary tract infection until appropriately treated
7. Participants with preexisting conditions, which, in the opinion of the investigator, interfere with the conduct of the study

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2025-04-16 (Estimated); Study Completion 2025-04-16 (Estimated)

PRIMARY OUTCOMES:
Comparison of Operating Time | Intra-op
  Operating time as measured during the procedure measured in minutes.

SECONDARY OUTCOMES:
Time to Catheter Removal | Within 6 hours of procedure completion
  Time from end of procedure to the removal of catheter measured in minutes.
Length of Hospital Stay | Within 6 hours of procedure completion
  Time from end of procedure to participant discharge from the hospital in minutes.
Continence status | One year post-procedure
  Self-report from the participant on their continence.
International Prostate Symptom Score | One year post-procedure
  Eight questions (seven concerning urinary symptoms and one concerning quality of life), responses range from 0 (better outcome) to 5 (worse outcome), with total score ranging from 0 to 35.
Quality of Life (QOL) as scored on the International Prostate Symptom Score (IPSS) | One year post-procedure
  Response to the last question on the IPSS:
  "If you were to spend the rest of your life with your urinary condition just the way it is now, how would you feel about that?" Response ranging from 'Delighted' to 'Terrible
Peak flow rate | One year post-procedure
  Measured as Qmax "If you were to spend the rest of your life with your urinary condition just the way it is now, how would you feel about that?" Response ranging from 'Delighted' to 'Terrible
Post-void residual | One year post-procedure
  PVR "If you were to spend the rest of your life with your urinary condition just the way it is now, how would you feel about that?" Response ranging from 'Delighted' to 'Terrible
Rate of Complications | One year post-procedure
  Occurrence of procedure-related complications

CONTACTS AND LOCATIONS:
Overall Officials: Hazem Elmansy, Principal Investigator — Thunder Bay Regional Health Sciences Centre
Locations (1):
- Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No